CLINICAL TRIAL: NCT06455202
Title: A Phase 3 Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy and Safety of Barzolvolimab in Patients With Chronic Spontaneous Urticaria Who Remain Symptomatic Despite H1 Antihistamine Treatment (EMBARQ-CSU2)
Brief Title: A Phase 3 Study of Barzolvolimab in Participants With Chronic Spontaneous Urticaria (CSU)
Acronym: EMBARQ-CSU2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Celldex Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CDX0159-13; 2024-513210-36-00 (EU CTIS Number)
Record Dates: First submitted 2024-06-07; First posted 2024-06-12 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Chronic Spontaneous Urticaria
Keywords: CDX-0159; barzolvolimab; chronic spontaneous urticaria; CSU; urticaria activity score; itch severity score; hives severity score
MeSH Terms: conditions — Chronic Urticaria

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- barzolvolimab 150 mg (Experimental): barzolvolimab given once as a 300 mg subcutaneous injection followed by 150 mg administered every 4 weeks for 52 weeks
  Interventions: Biological: barzolvolimab
- barzolvolimab 300 mg (Experimental): barzolvolimab given once as a 450 mg subcutaneous injection followed by 300 mg administered every 8 weeks for 52 weeks
  Interventions: Biological: barzolvolimab
- Placebo then barzolvolimab 150 mg (Experimental): Placebo injection subcutaneous every 4 weeks for 24 weeks and then barzolvolimab 300 mg followed by 150 mg administered every 4 weeks for 28 weeks.
  Interventions: Biological: barzolvolimab; Biological: Matching placebo
- Placebo then barzolvolimab 300 mg (Experimental): Placebo injection subcutaneous every 4 weeks for 24 weeks and then barzolvolimab 450 mg followed by 300 mg administered every 8 weeks for 28 weeks.
  Interventions: Biological: barzolvolimab; Biological: Matching placebo

INTERVENTIONS:
Biological: barzolvolimab — Subcutaneous Administration
Biological: Matching placebo — Matching placebo Subcutaneous Administration
  Arms: Placebo then barzolvolimab 150 mg; Placebo then barzolvolimab 300 mg

SUMMARY:
The purpose of this study is to establish the efficacy, safety and tolerability of barzolvolimab in adult participants with Chronic Spontaneous Urticaria (CSU) inadequately controlled by non-sedating second generation H1-antihistamines in comparison to placebo.

DETAILED DESCRIPTION:
This is a global, multicenter, randomized, double-blind, parallel group, placebo-controlled phase 3 study investigating the efficacy, safety and tolerability of barzolvolimab in adult participants with Chronic Spontaneous Urticaria (CSU) who are symptomatic despite treatment with non-sedating second generation H1-antihistamines at 1-4 times the locally approved dose.

There is a screening period of up to 4 weeks, followed by a 24-week placebo-controlled treatment period, a 28-week active treatment period where all participants receive barzolvolimab followed by a 16-week treatment free period.

Approximately 915 adult participants (610 in the active arms and 305 in the placebo arm) will be randomly assigned to the treatment arms.

ELIGIBILITY:
Key Inclusion Criteria:

1. Males and females, >/= 18 years of age.
2. Chronic spontaneous urticaria (CSU) >/= 6 months prior to Screening (Visit 1).
3. CSU despite the use of a stable regimen of second generation non-sedating H1-antihistamine as defined by:

   1. The presence of hives for >/= 6 weeks at any time prior to Visit 1 despite the use of non-sedating H1-antihistamines.
   2. Must be on a stable regimen of second generation non-sedating H1-antihistamine for >/= 4 weeks prior to study treatment.
   3. UAS7 of >/= 16 and ISS7 of >/= 8 during the 7 days prior to study treatment.
4. Normal blood counts and liver function tests.
5. Both males and females of child-bearing potential must agree to use highly effective contraceptives during the study and for 150 days after treatment.
6. Willing and able to complete a daily symptom electronic diary and comply with study visits.
7. Participants with and without prior biologic experience are eligible.

Key Exclusion Criteria:

1. Women who are pregnant or nursing.
2. Chronic urticaria whose predominant manifestation is due to CIndU.
3. Other diseases associated with urticaria.
4. Active pruritic skin condition in addition to CSU.
5. Medical condition that would cause additional risk or interfere with study procedures.
6. Known HIV, hepatitis B or hepatitis C infection.
7. Vaccination of a live vaccine within 30 days prior to Screening (Visit 1) (subjects must agree to avoid live vaccinations during the study). Inactivated vaccines are allowed such as seasonal influenza injection or authorized COVID-19 vaccine.
8. History of anaphylaxis
9. Prior treatment with barzolvolimab

There are additional criteria that your study doctor will review with you to confirm you are eligible for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 915 (Estimated)
Dates: Start 2024-07-19 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline to Week 12 of UAS7 (Urticaria Activity Score) | From Day 1 (first dose) to Day 85 (Week 12)
  Evaluate efficacy of barzolvolimab on urticaria activity as measured by urticaria activity score (UAS).
  The UAS7 is a simple scoring system to evaluate urticaria signs and symptoms. It is based on scoring wheals (hive severity score) and itch (itch severity score) separately on a scale of 0 (no signs/symptoms) to 3 (intense signs/symptoms) over 7 days. The final score is calculated by adding together the daily scores, which can range from 0 to 6, for 7 days. This results in a maximum total score of 42, and a minimum possible score of 0.

SECONDARY OUTCOMES:
Mean change from baseline to Week 12 of ISS7 (Itch Severity Score) | From Day 1 (first dose) to Day 85 (Week 12)
  The ISS7 and HSS7 combined together make up the UAS7 scoring system to evaluate urticaria signs and symptoms. The ISS7 is the itch severity score for 7 days, the scores range from 0 to 21.
Mean change from baseline to Week 12 of HSS7 (Hives Severity Score) | From Day 1 (first dose) to Day 85 (Week 12)
  The ISS7 and HSS7 combined together make up the UAS7 scoring system to evaluate urticaria signs and symptoms. The HSS7 score is the wheal/hives severity score for 7 days, the scores range from 0 to 21.
Percentage of patients with UAS7=0 at Week 12 | From Day 1 (first dose) to Day 85 (Week 12)
  Proportion of participants who achieve complete absence of hives and itch (UAS7 = 0) at Week 12.
Percentage of participants with UAS7 ≤ 6 at Week 12 | From Day 1 (first dose) to Day 85 (Week 12)
  Proportion of participants who achieve control of their urticaria signs and symptoms (UAS7≤6) at Week 12.
Percentage of participants with AAS7 > 0 at baseline with AAS7 = 0 at Week 12 | From Day 1 (first dose) to Day 85 (Week 12)
  Proportion of participants with AAS7 > 0 at Day 1 who achieved complete control (AAS7 = 0) at Week 12
  Angioedema Activity Score over 7 days [AAS7] describes the effect of angioedema on five categories with 0 being none and 3 being most severe. The final score is calculated by adding together daily scores which can range from 0-15 for 7 days. The resulting maximum score is then 105.
Mean change from baseline in UAS7 in participants refractory to omalizumab treatment at Week 12 | From Day 1 (first dose) to Day 85 (Week 12)
  Evaluate efficacy of barzolvolimab on urticaria activity as measured by urticaria activity score (UAS) in participants who did not respond to or did not tolerate omalizumab.
  The UAS7 is a simple scoring system to evaluate urticaria signs and symptoms. It is based on scoring wheals (hive severity score) and itch (itch severity score) separately on a scale of 0 (no signs/symptoms) to 3 (intense signs/symptoms) over 7 days. The final score is calculated by adding together the daily scores, which can range from 0 to 6, for 7 days. This results in a maximum total score of 42, and a minimum possible score of 0.
Proportion of participants with UAS7 = 0 in participants refractory to omalizumab treatment at Week 12 | From Day 1 (first dose) to Day 85 (Week 12)
  Proportion of participants who achieve complete absence of hives and itch (UAS7 = 0) at Week 12 in participants who did not respond to or did not tolerate omalizumab.
Incidence of Treatment-Emergent Adverse Events | From Day 1 (first dose) to Day 477 (Week 68)
  Occurrence of treatment emergent adverse events and serious adverse events during the study.

CONTACTS AND LOCATIONS:
Locations (260):
- United States (71):
  - Allervie Clinical Research - Cullman, Cullman, Alabama
  - Research Solutions of Arizona PC, Litchfield Park, Arizona
  - Medical Research of Arizona a division of Allergy, Asthma, & Immunology, Assoc. Ltd., Scottsdale, Arizona
  - Center for Dermatology & Plastic Surgery, Scottsdale, Arizona
  - Burke Pharmaceutical Research, Hot Springs, Arkansas
  - Kern Research, Inc., Bakersfield, California
  - UCLA Clinical Trials Contracts & Strategic Relations, Los Angeles, California
  - California Allergy and Asthma Medical Group, Los Angeles, California
  - LA Universal Research Center, Inc., Los Angeles, California
  - Allergy and Asthma Associates of Southern Cal, Mission Viejo, California
  - Huntington Asthma & Allergy Center, Pasadena, California
  - Apex Clinical Research, San Diego, California
  - WR-MCCR, San Diego, California
  - University Clinical Trials, San Diego, California
  - Clinical Science Institute, Santa Monica, California
  - Raffi Tachdjian MD, Inc, Santa Monica, California
  - Clarity Dermatology, PLLC, Castle Rock, Colorado
  - Asthma and Allergy Associates, Colorado Springs, Colorado
  - ClearlyDerm Boca Raton - ClinEdge - PPDS, Boca Raton, Florida
  - Driven Research LLC, Coral Gables, Florida
  - Palm Beach Dermatology Group, Delray Beach, Florida
  - Dolphin Medical Research, Doral, Florida
  - South FL Clinical Research LLC, Miami, Florida
  - Dade Florida Clinical Research Center, Miami, Florida
  - Deluxe Health Center, Miami Lakes, Florida
  - Revival Clinical Research, Orlando, Florida
  - International Clinical Research - FL LLC, Sanford, Florida
  - Allergy and Asthma Diagnostic treatment Center - CRN - PPDS, Tallahassee, Florida
  - D&H Tamarac Research Center, LLC, Tamarac, Florida
  - Advanced Clinical Research Institute (ACRI) - Florida, Tampa, Florida
  - Deluxe Health Center, Tampa, Florida
  - MOORE Clinical Research, Inc. d/b/a TrueBlue Clinical Research, Tampa, Florida
  - University of South Florida, Tampa, Florida
  - Olympian Clinical Research, Tampa, Florida
  - Lane Dermatology Research - Centricity - PPDS, Columbus, Georgia
  - Skin Care Physicians of Georgia, Macon, Georgia
  - Treasure Valley Medical Research, Boise, Idaho
  - Rush University Medical Center, Chicago, Illinois
  - Sneeze Wheeze and Itch Associates LLC, Normal, Illinois
  - The Indiana Clinical Trials Center, PC, Plainfield, Indiana
  - South Bend Clinic, South Bend, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Henry J. Kanarek - Allergy,Asthma&Immunology, Overland Park, Kansas
  - Equity Medical, Bowling Green, Kentucky
  - Allergy & Asthma Associates, Lexington, Kentucky
  - Velocity Clinical Research - The Dermatology Clinic - Baton Rouge - PPDS, Baton Rouge, Louisiana
  - Continental Clinical Research Solutions, LLC - ClinEdge - PPDS, Towson, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Derm Institute of Western Michigan, Caledonia, Michigan
  - Clarkston Skin Research - Clarkston, Clarkston, Michigan
  - Grekin Skin Institute, Warren, Michigan
  - Midwest Clinical Research, LLC, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Skin Specialists PC, Omaha, Nebraska
  - Hudson-Essex Allergy, Belleville, New Jersey
  - Impact Medical / Circuit Clinical, Paramus, New Jersey
  - Impact Medical / Circuit Clinical, Riverdale, New Jersey
  - Equity Medical LLC, New York, New York
  - OptiSkin Medical, New York, New York
  - Optima Research, Boardman, Ohio
  - Optimed Research Ltd - ClinEdge - PPDS, Columbus, Ohio
  - Penn State Health Milton Hershey Med Cen, Hershey, Pennsylvania
  - Clinical Partners LLC, Johnston, Rhode Island
  - University of Texas Health McGovern Medical, Bellaire, Texas
  - Western Sky Medical Research, El Paso, Texas
  - Austin Institute for Clinical Research, Inc., Pflugerville, Texas
  - Rainey & Finklea San Antonio Dermatology, San Antonio, Texas
  - Allergy Associates of Utah - Sandy, Murray, Utah
  - Jordan Valley Dermatology Center-South Jordan, South Jordan, Utah
  - Kalo Clinical Research, West Valley City, Utah
  - Virginia Dermatology and Skin Cancer Center - Norfolk, Norfolk, Virginia
- Australia (12):
  - Novatrials, Charlestown, New South Wales
  - Skin and Cancer Foundation - The Skin Hospital, Darlinghurst, New South Wales
  - St George Dermatology and Skin Cancer Center, Kogarah, New South Wales
  - Momentum Clinical Research Darlinghurst, Sydney, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Cornerstone Dermatology, Coorparoo, Queensland
  - Veracity Clinical Research Pty Ltd, Woolloongabba, Queensland
  - Box Hill Hospital, Box Hill, Victoria
  - Dr Rodney Sinclair Pty Ltd, East Melbourne, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - The Royal Melbourne Hospital, Parkville, Victoria
- Bulgaria (12):
  - Medical Centre Asklepii OOD, Dupnitsa
  - Medical Center - Pulmo 2018, Haskovo
  - Medical Center Medconsult Pleven, Lovech
  - Multiprofile Hospital for Active Treatment - Pazardzhik AD, Pazardzhik
  - University Multiprofile Hospital for Active Treatment Sveti Georgi EAD, Plovdiv
  - Medical Center Prolet, Rousse
  - Medical Center Unimed EOOD, Sevlievo
  - Diagnostic-consultative center Ascendent EOOD, Sofia
  - Diagnostic and Consultative Center Aleksandrovska EOOD, Sofia
  - University Multiprofile Hospital for Active Treatment Aleksandrovska EAD, Sofia
  - University Multiprofile Hospital for Active Treatment "Tsaritsa Yoanna - ISUL", Sofia
  - Diagnostic-Consultative Centre Convex EOOD, Sofia
- Canada (13):
  - Laser Rejuvenation Clinics Edmonton D.T. Inc., Edmonton, Alberta
  - Vida Clinical Research, Edmonton, Alberta
  - Rejuvenation Dermatology Edmonton South, Edmonton, Alberta
  - LEADER research, Hamilton, Ontario
  - DermEffects, London, Ontario
  - North Bay Dermatology Centre, North Bay, Ontario
  - Ottawa Allergy Research Corporation, Ottawa, Ontario
  - York Dermatology Clinic & Research Centre, Richmond Hill, Ontario
  - North York Research Inc., Toronto, Ontario
  - Joel Liem Medicine Professional Corporation, Windsor, Ontario
  - Saskatoon Dermatology Centre, Saskatoon, Saskatchewan
  - Kingston Health Science Center, Kingston
  - Centre de Recherche Saint-Louis (Québec), Québec
- Chile (8):
  - Clinica MEDS La Dehesa, Lo Barnechea
  - Hospital Base San Jose de Osorno, Osorno
  - Enroll SpA - Dr. Manuel Barros Borgono, Providencia
  - Clinica Davila - Recoleta, Recoleta
  - Centro Internacional de Estudios Clinicos (CIEC), Recoleta
  - BIOCINETIC Ltda, Santiago
  - Medical Skin Center, Viña del Mar
  - Dermacross Clinica Dermatologica, Vitacura
- Colombia (6):
  - Centro Integral de Reumatologia Del Caribe, Barranquilla
  - Hospital Alma Mater de Antioquia, Medellín
  - Centro de Inmunología y Genética - CIGE S.A.S, Medellín
  - Hospital General de Medellín Luz Castro de Gutiérrez, Medellín
  - Fundación Centro de Investigation Clínica CIC, Medellín
  - Fundación Hospital Universidad del Norte, Soledad
- Croatia (2):
  - Special Hospital Medico, Rijeka
  - Solmed Clinic, Zagreb
- Georgia (4):
  - LTD" Healthy Future", Tbilisi
  - LTD "Center of Allergy and Immunology", Tbilisi
  - David Abuladze Georgian Italian Clinic, Tbilisi
  - LTD "Multiprofile Clinic Consilium Medulla", Tbilisi
- Germany (14):
  - Universitätsklinikum der RWTH Aachen Hautklinik, Aachen
  - Fachklinik Bad Bentheim, Bad Bentheim
  - Emovis GmbH, Berlin
  - Universitätsklinikum Bonn, Bonn
  - Klinische Forschung Dresden GmbH, Dresden
  - Universitätsklinikum Carl Gustav Carus an der TU Dresden, Dresden
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Universitätsklinikum Essen, Essen
  - Eurofins bioskin Research Center Dermalology, Hamburg
  - UKSH Lübeck, Institut für Entzündungsmedizin, Lübeck
  - Universitätsklinikum Mannheim, Mannheim
  - Universitätsklinikum Münster, Münster
  - Hautarztpraxis Dariusch Mortazawi, Remscheid
  - Universitäts-Hautklinik, Studienzentrum Immundermatologie, Tübingen
- Hungary (3):
  - Debreceni Egyetem Klinikai Kozpont Nagyerdei Campus, Debrecen
  - Szent-Gyorgyi Albert Klinikai Kozpont, Szeged
  - Allergo-Derm Bakos Kft., Szolnok
- India (15):
  - Nirmal Hospital PVT LTD, Surat, Gujarat
  - Medical College Baroda & SSG Hospital, Vadodara, Gujarat
  - Shree Hospital & Critical Care Centre, Nagpur, Maharashtra
  - Assured Care Plus Hospital, Nashik, Maharashtra
  - Oyster & Pearl Hospitals, Pune, Maharashtra
  - Excelcare Hospital, Jaipur, Rajasthan
  - G.S.V.M. Medical College - Kanpur, Kanpur, Uttar Pradesh
  - Panchshil Hospital - Ahmedabad, Ahmedabad
  - B. J. Medical College and Civil Hospital, Ahmedabad
  - KLES Dr Prabhakar Kore Hospital & Medical Research Centre, Belagavi
  - All India Institute of Medical Sciences, Bhubaneswar
  - Apex Hospitals Pvt Ltd, Jaipur
  - K R Hospital, Mysore
  - Deenanath Mangeshkar Hospital and Research Centre, Pune
  - Sumandeep Vidyapeeth University - Dhiraj Hospital, Vadodara
- Italy (7):
  - IRCCS Ospedale Policlinico San Martino, Genova
  - Asst Fbf Sacco, Milan
  - Azienda Ospedale Università di Padova, Padua
  - Humanitas Research Hospital, Rozzano
  - AOU San Giovanni di Dio e Ruggi d'Aragona, Salerno
  - IRCCS Policlinico San Donato, San Donato Milanese
  - Ospedale San Lazzaro PO Molinette, Torino
- Lithuania (4):
  - CD8 Klinika, Kaunas
  - UAB Ausros Medicinos Centras, Kaunas
  - UAB "Alerginių susirgimų diagnostikos ir gydymo centras", Vilnius
  - Santaros KTC (klinikiniu tyrimu centras), Vilnius
- Mexico (12):
  - Unidad de Investigación Cima S.a, Chihuahua City
  - Meidadvance Clinical, Chihuahua City
  - Cryptex, Cuauhtémoc
  - Centro de Investigación Medico Biologica, Guadalajara
  - CIMET, Guadalajara
  - Panamerican Guadalajara, Guadalajara
  - Centro de Desarrollo Biomédico, Mérida
  - Mérida Investigación Clínica, Mérida
  - Eukarya Pharmasite, Monterrey
  - CECYPE, Morelia
  - Unidad de Medicina Especializada, San Juan del Río
  - FAICIC, Veracruz
- Netherlands (3):
  - AmdsterdamUMC locatie AMC, Amsterdam
  - Bravis Hospital, Roosendaal
  - University Medical Center Utrecht, Utrecht
- New Zealand (8):
  - Optimal Clinical Trials - Central, Auckland
  - Pcrn Chch, Christchurch
  - Momentum Clinical Research Dunedin, Dunedin
  - Lakeland Clinical Trials - Waikato, Hamilton
  - velocity Nova Sp. z o.o., Nelson
  - Pacific Clinical Research Network Rotorua, Rotorua
  - Momentum Clinical Research Tauranga, Tauranga
  - Lakeland Clinical Trials Wellington, Upper Hutt
- Poland (26):
  - Klinika Dermatologii i Dermatologii Onkologicznej, Częstochowa
  - Centrum Medyczne Pratia Częstochowa, Częstochowa
  - Centrum Kliniczno-Badawcze J.Brzezicki,B.Górnikiewicz-Brzezicka, Lekarze Spółka Partnerska, Elblag
  - Synexus Polska Sp. z o.o., Gdansk
  - Mazowieckie Centrum Badań Klinicznych SC IWONA CZAJKOWSKA ANNA PODRAZKA-SZCZEAPANIAK, Grodzisk Mazowiecki
  - Provita Sp zoo, Katowice
  - Centrum Medyczne "All-Med" Badania Kliniczne, Krakow
  - Centrum Medyczne Plejady, Krakow
  - Malopolskie Centrum Alergologii, Krakow
  - Uniwersytet Medyczny w Łodzi - Centrum Wsparcia Badań Klinicznych, Lodz
  - Velocity Nova Sp. z o.o., Lublin
  - Pro Life Medica ETG Lublin, Lublin
  - DERMEDIC Iwona Zdybska, Lublin
  - LUXDERM Specjalistyczny Gabinet Dermatologiczny Prof. dr hab. n. med. Dorota Krasowska, Lublin
  - Twoja Przychodnia Nowosolskie Centrum Medyczne, Nowa Sól
  - Uniwersytecki Szpital Kliniczny w Opolu, Opole
  - Medicome Sp. Z O.O., Oświęcim
  - Centrum Alergologii Teresa Hofman Sp. z.o.o., Poznan
  - EMC Instytut Medyczny SA, PL Certus Szpital i Ambulatorium, Poznan
  - Specjalistyczny Niepubliczny Zaklad Opieki Zdrowotnej Alergologia Plus Osrodek Diagnostyki I Terapii Uczulen, Poznan
  - Uniwersytecki Szpital Kliniczny im. Fryderka Chopina w Rzeszowie Klinika Dermatologii i Dermatologii Onkologicznej, Rzeszów
  - EMED Centrum Usług Medycznych Ewa Śmiałek, Rzeszów
  - ALERGO-MED SPECJALISTYCZNA PRZYCHODNIA LEKARSKA Spolka. z o. o., Tarnów
  - Medicover Integrated Clinical Services Sp. z o.o. Centrum Medyczne Warszawa, Warsaw
  - Synexus Polska Sp. z o.o., Warsaw
  - ETG Warszawa, Warsaw
- Slovakia (5):
  - MAXDERM s.r.o., Bardejov
  - Cliniq s.r.o., Bratislava
  - Derma therapy spol. s.r.o., Bratislava
  - ALERSA, sro, Košice
  - Fakultna nemocnica Trnava, Trnava
- Spain (14):
  - Hospital del Mar, Barcelona
  - Hospital Universitari Puerta del Mar, Cadiz
  - Hospital Universitario de La Princesa, Madrid
  - Clinica Universidad Navarra- Madrid, Madrid
  - Hospital 12 De Octubre, Madrid
  - Hospital Universitario Fundación Alcorcón, Madrid
  - Clinica Universidad Navarra- Pamplona, Pamplona
  - Complejo Hospitalario Universitario de Pontevedra- Centro Especialidades de Mollabao, Pontevedra
  - Hospital Quironsalud Madrid, Pozuelo de Alarcón
  - Hospital universitario Virgen Macarena, Seville
  - FutureMeds Sevilla, Seville
  - Hospital Universitario de Torrejón, Torrejón de Ardoz
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
  - Hospital de Manises, Valencia
- Thailand (4):
  - Siriraj Hospital, Bangkok Noi
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai
  - Thammasat University Hospital, Khlong Luang
  - Khon Kaen University, Khon Kaen
- Tunisia (3):
  - Hôpital Hédi Chaker, Sfax
  - La Rabta Hospital, Tunis
  - Habib Thameur Hospital, Tunis
- United Kingdom (14):
  - Southmead Hospital, Bristol
  - Velocity Clinical Research - Bristol, Bristol
  - Cambridge University Hospitals, Addenbrooke's Hospital, Cambridge
  - Western General Hospital, Edinburgh
  - Queen Elizabeth University Hospital, Glasgow
  - Velocity Clinical Research High Wycombe, High Wycombe
  - St James's University Hospital, Leeds
  - The Royal London Hospital, London
  - Velocity Clinical Research, North London - PPDS, North Finchley
  - Virtual Clinical Trials Centre, The Stables, Oxford
  - University Hospitals Plymouth NHS Trust, Plymouth
  - Royal Berkshire Hospital, Reading
  - Velocity Clinical Research - Romford, Romford
  - Pinderfields Hospital, Wakefield

IPD SHARING:
Plan to Share IPD: Undecided